CLINICAL TRIAL: NCT06770465
Title: Maternal Use of Antibiotics and the Risk of Congenital Malformations: a Study Using Spontaneous Reporting Data and a Population-based Cohort Data From the US, Canada and China
Brief Title: Maternal Use of Antibiotics and the Risk of Congenital Malformations
Status: Active, not recruiting | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Sun Xin, professor, West China Hospital
Other Study IDs: Antibiotics and BDs
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Congenital Malformations
Keywords: Antibiotic; Congenital malformation; Pregnancy; Spontaneous report; Cohort
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Use of antibiotics during pregnancy in FAERS and CVAR databases: When using the publicly available spontaneous adverse event reporting databases FAERS and CVAR, the exposure group consists of reports of adverse events in pregnant individuals who used different types of antibiotics, and the control group consists of other adverse event reports in which no antibiotics were used.
  Interventions: Drug: Different categories of antibiotics
- Use of antibiotics during pregnancy in a cohort in Xiamen, China: When using the pregnant women cohort data from Xiamen, China, the exposure group consists of pregnant individuals who used the target antibiotics of interest, while the control group is either those who did not use any antibiotics (blank control) or those who used penicillin (positive control).
  Interventions: Drug: Different categories of antibiotics

INTERVENTIONS:
Drug: Different categories of antibiotics — Use of different categories of antibiotics during pregnancy, such as quinolones and macrolides.

SUMMARY:
Antibiotics are widely used during pregnancy to prevent or treat infections, yet concerns remain regarding their fetal safety. Drawing on data from spontaneous reporting databases and cohort studies, this study aims to explore potential associations between exposure to various antibiotic classes during pregnancy and congenital malformations.

Data were collected from publicly available reports in the U.S. Food and Drug Administration's Adverse Event Reporting System (FAERS), the Canada Vigilance Adverse Reaction (CVAR) database, and a population-based retrospective cohort in Xiamen, China. By applying multiple signal detection methods, we identified potential risk signals linking different antibiotic classes to organ-system-specific congenital malformations. For antibiotics showing positive signals, we further utilized a pregnancy medication cohort in Xiamen and applied causal inference techniques to estimate the adjusted relative risk of congenital malformations associated with first-trimester exposure to these antibiotics. Several sensitivity analyses-including both negative- and positive-control analyses-will also be performed.

ELIGIBILITY:
Inclusion Criteria:

* For the spontaneous reporting data study, all adverse reactions reported by mothers were included.

For the cohort study, all Xiamen pregnant women registered in the cohort were included

Exclusion Criteria:

* For studies using spontaneous reporting data, all adverse reaction reports unrelated to pregnant or postpartum women-including those occurring during the lactation period-were excluded.

For cohort studies, pregnant women who were lost to follow-up were excluded, and pregnant women who were exposed to factors known to be associated with congenital malformations were excluded.

Ages: 14 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: For the spontaneous reporting studies, the study population was pregnant women who reported an adverse medication event during the study period, where the exposed population was pregnant women who reported an adverse event due to the use of a different type of antibiotic during the study period.
  For cohort studies, the study population was women who were pregnant during the study period and the exposed population was pregnant women who used different types of antibiotics during the study period
Sampling Method: Non-Probability Sample
Enrollment: 850000 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Congenital malformations | From pregnancy to 42 days after delivery
  This study categorizes congenital malformation adverse events into 10 organ system specific congenital malformation (Q00-Q89) based on ICQ-10. Additionally, the cohort detected 22 congenital malformations mandated for surveillance in China and generated a composite outcome of total congenital malformation, that was a combination of all the above congenital anomalies.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Sun, PhD, Study Chair — Chinese Evidence-based Medicine Center, West China Hospital of Sichuan University
Locations (1):
- The West China Hospital of Sichuan university, Chengdu, Sichuan, China